CLINICAL TRIAL: NCT05827666
Title: The Effect of Dairy and Dairy-Free Alternative Beverages on Post-Exercise Anabolism in Active Youth
Acronym: PBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Collaborators: Dairy Management Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 43728
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Dietary Proteins; Indicator Amino Acid Oxidation
Keywords: Nutrition in Youth; Growth; Active youth; Protein metabolism; Lean body mass; Whole food matrix; Protein beverage; Children; Adolescent; Indicator Amino Acid Oxidation
MeSH Terms: interventions — Milk

STUDY DESIGN:
Intervention Model Description: Using a single-blind randomized counterbalanced crossover design, participants will complete four metabolic trials providing one of the four isoenergetic (equal calories) beverages: 2% milk (MILK), soy 'milk,' (SOY), almond 'milk,' (ALMOND), or rice 'milk' (RICE) following a bout of variable-intensity exercise. The caloric content of the beverages is based on 0.3 g/kg FFM 2% milk.
Who Masked: Participant
Masking Description: As the study is a single-blind crossover design, the randomization of the protein type will be blinded to the participants only. For each liquid meal, beverages will be provided in opaque bottles, and the caloric content of the beverages will be the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children (Active Comparator): Participants will undergo four metabolic trials in a randomized crossover design, where they will be provided with an isoenergetic (i.e., equal calories) amount of one of the following beverages upon completing a standardized bout of variably intensity exercise: 2% milk, almond 'milk,' soy 'milk,' or rice 'milk.'
  Interventions: Dietary Supplement: 2% milk beverage; Dietary Supplement: Almond milk alternative beverage; Dietary Supplement: Soy milk alternative beverage; Dietary Supplement: Rice milk alternative beverage
- Adolescent females (Active Comparator): Participants will undergo four metabolic trials in a randomized crossover design, where they will be provided with an isoenergetic (i.e., equal calories) amount of one of the following beverages upon completing a standardized bout of variably intensity exercise: 2% milk, almond 'milk,' soy 'milk,' or rice 'milk.'
  Interventions: Dietary Supplement: 2% milk beverage; Dietary Supplement: Almond milk alternative beverage; Dietary Supplement: Soy milk alternative beverage; Dietary Supplement: Rice milk alternative beverage
- Adolescent males (Active Comparator): Participants will undergo four metabolic trials in a randomized crossover design, where they will be provided with an isoenergetic (i.e., equal calories) amount of one of the following beverages upon completing a standardized bout of variably intensity exercise: 2% milk, almond 'milk,' soy 'milk,' or rice 'milk.'
  Interventions: Dietary Supplement: 2% milk beverage; Dietary Supplement: Almond milk alternative beverage; Dietary Supplement: Soy milk alternative beverage; Dietary Supplement: Rice milk alternative beverage

INTERVENTIONS:
Dietary Supplement: 2% milk beverage — Protein provided at 0.3 g/kg fat-free mass. All other conditions (almond, soy and rice milk alternative beverages) will be matched to the same energy content (i.e., isoenergetic). Macronutrient content of beverage (per 100 g): Calories: 52 kcal; Fat: 2.25 g; Carbohydrates: 4.8 g; Protein: 3.3 g.
  Other Names: Natrel 2% milk
Dietary Supplement: Almond milk alternative beverage — Matched to the same energy intake as 0.3 g/kg FFM of 2% milk. Macronutrient content of beverage (per 100 g): Calories: 24 kcal; Fat: 1.13 g; Carbohydrates: 3.1 g; Protein: 0.3 g.
  Other Names: Silk Original Almond Beverage
Dietary Supplement: Soy milk alternative beverage — Matched to the same energy intake as 0.3 g/kg FFM of 2% milk. Macronutrient content of beverage (per 100 g): Calories: 39 kcal; Fat: 1.70 g; Carbohydrates: 3.0 g; Protein: 2.9 g.
  Other Names: Silk Original Soy Beverage
Dietary Supplement: Rice milk alternative beverage — Matched to the same energy intake as 0.3 g/kg FFM of 2% milk. Macronutrient content of beverage (per 100 g): Calories: 49 kcal; Fat: 1.09 g; Carbohydrates: 9.8 g; Protein: 0.1 g.
  Other Names: Rice Dream Milk Beverage

SUMMARY:
The growth and development of lean body mass (i.e., muscle and bone) is instrumental to health and performance across the lifespan, especially in youth, as they actively experience growth. Thus, it is important to capitalize on physical activity and nutrition (especially dietary protein), to support the accretion of lean tissues. Eating a protein-rich meal or performing physical activity can stimulate protein synthesis, and when repeated over time, lean body mass accretion. There is currently an increasing market demand for non-dairy alternatives, due to multiple reasons including environmental, ethical, or taste preferences. However, it is important to understand how different beverages may support 'growth' (anabolism) of lean tissues after exercise. Research in adults has shown that dairy milk is superior to non-dairy milk beverages for supporting post-exercise recovery and muscle protein synthesis. However, the impact of dairy and non-dairy milk alternatives on recovery from exercise is not well understood in children. By understanding the milk beverage that best supports post-exercise recovery, the investigators can determine the optimal nutritional environment to facilitate the growth of lean tissues in the body.

DETAILED DESCRIPTION:
The growth and development of lean body mass (LBM) (e.g., muscle and bone) is vital to not only support health and performance across the lifespan but also, reduce the prevalence of metabolic disorders later in life, such as osteoporosis and sarcopenia. Active youth who regularly perform moderate-to-vigorous physical activity (MVPA) have superior increases LBM and muscle strength compared to their sedentary counterparts. LBM is regulated by the process of protein breakdown (PB), where old or damaged proteins are broken down releasing their constituent amino acids (AA), as well as protein synthesis (PS), a process by which new proteins are made by linking constituent AAs together. When rates of PS exceed rates of PB (PS>PB), a positive net protein balance is achieved, ultimately facilitating the accretion of LBM. Contrarily, if PB>PS, net protein balance is negative, leading to the loss of LBM.

Assuming total energy intakes are met, to meet the metabolic demands of an active lifestyle, dietary protein is a prime anabolic stimulus. This macronutrient facilitates the growth of lean tissues by providing the AA 'building blocks' to support the synthesis of muscle and other body proteins. Physical activity (PA) is a second pre-eminent factor contributing to the growth of LBM. Following exercise, in the absence of dietary protein ingestion, net protein balance is negative. However, post-exercise protein consumption facilitates a positive net protein balance, which when repeated over time, can contribute to the accretion of LBM. Youth who engage in high levels of PA have greater LBM compared to their sedentary counterparts. Thus, it is important to capitalize on the optimal nutritional and exercise interventions to support a positive net protein balance, an acute marker of growth, especially in vulnerable populations, such as children.

In children, milk protein ingestion has been shown to stimulate whole-body PS, resulting in a positive whole-body net protein balance. In adults, dairy proteins lead to superior post-exercise recovery and PS compared to non-dairy alternatives. Most research to date examining the post-prandial protein synthesis responses to plant-based protein sources have encompassed isolated protein sources. However, there is currently a paucity of research examining the effect of the whole-food matrix of plant-based protein sources on whole-body protein metabolism in active youth. Furthermore, the pubertal growth spurt is characterized by rapid accumulation of LBM that is only surpassed by the first year of life. This LBM, which is enhanced by an active lifestyle, must be supported by adequate energy and protein ingestion. Therefore, it is necessary to determine the post-exercise anabolic effect of dairy and non-dairy whole foods on markers of LBM growth and whole-body protein metabolism, especially in children, an under-researched population.

The current project will employ the indicator amino acid oxidation (IAAO) methodology to determine the protein/AA intake that minimizes oxidation of the indicator AA, while maximizing PS. The oxidation of the indicator AA is minimized by ingesting an adequate proportion of AA, and/or consuming nutritionally complete protein sources. The main objective of the present study is to determine the effect of energy-matched dairy and non-dairy milk alternatives on whole-body protein synthesis in active youth following exercise.

Aim 1: To determine the effect of dairy (2% milk) and non-dairy milk alternatives (soy, rice, and almond 'milk' beverages) on whole-body PS following a bout of intermittent exercise in children, adolescent males, and adolescent females.

Hypothesis 1: Whole body PS will be greatest after ingestion of dairy milk compared to isocaloric (i.e., equal energy amount) non-dairy alternatives, due to the greater and/or higher amount of quality dietary protein. Regardless of sex, adolescents are expected to have greater PS due to their heightened anabolic sensitivity, compared to children.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 8-16 years
* Children: >-1 y age from peak height velocity* (aPHV)
* Adolescents: -0.5 to 1.5 aPHV
* An age and sex-specific minimum of 75th percentile Beep Test level
* Considered healthy based on responses to the PAR-Q+ and a medical history form *NOTE: age from peak height velocity (aPHV): sitting/standing height

Exclusion Criteria:

* Almond or soy allergy
* Lactose intolerance
* If enrolled as a child participant: biological age outside of >-1 years from aPHV
* If enrolled as an adolescent participant: biological age outside -0.5 to 1.5 aPHV
* Inability to perform physical activity as determined by the PAR-Q+ and iPAQ
* Inability to adhere to protocol guidelines (e.g., 2-day controlled diet)
* Diagnosed medical condition under the care of a physician (e.g., type 1 diabetes)
* Consuming any medications known to affect protein metabolism (e.g., corticosteroids, non-steroidal anti-inflammatories)
* Failure to complete all four metabolic trials within four months

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
F13CO2 | Duration of the metabolic trial (7 hours)
  The rate of 13CO2 excretion based upon baseline (t=30 minutes) and isotopic steady state (t=360-420 minutes) 13CO2 enrichments in the breath and resting VCO2

SECONDARY OUTCOMES:
Whole-Body Net Protein Balance | Duration of the metabolic trial (7 hours)
  Whole-Body Net Protein Balance will be calculated based upon baseline (t=30 minutes) and isotopic steady state (t=360-420 minutes) 13CO2 enrichments in the breath and 1-[13C]phenylalanine enrichments in the urine]

CONTACTS AND LOCATIONS:
Overall Officials: Nicki Pourhashemi, BSc, Study Director — University of Toronto
Locations (1):
- Goldring Centre for High Performance and Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No